CLINICAL TRIAL: NCT06895070
Title: PRESERVE CAP: A Prospective, Multi-Center, Single-Arm, Open-Label Study of Hearts Transplanted After Non-Ischemic Heart Preservation From Extended Donors Continued Access Protocol
Brief Title: XVIVO Heart Box (XHB) With Supplemented XVIVO Heart Solution (SXHS) Continued Access Protocol (CAP)
Acronym: NIHP-CAP-001
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XVIVO Perfusion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIHP-CAP-001
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-10

CONDITIONS: Heart Transplant; Heart Failure; Transplant; Failure, Heart
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Device: Preservation of hearts for transplant. (Experimental): Device: Preservation of hearts for transplant.
  Interventions: Device: Non-Ischemic Heart Preservation (NIHP) using the XVIVO Heart Assist Transport (XHAT)

INTERVENTIONS:
Device: Non-Ischemic Heart Preservation (NIHP) using the XVIVO Heart Assist Transport (XHAT) — Study donor hearts meeting extended criteria are preserved via Non-Ischemic Heart Preservation (NIHP) using the XVIVO Heart Preservation System (XHPS)

SUMMARY:
The purpose of this study is to evaluate if Non-Ischemic Heart Preservation (NIHP) of extended criteria donor hearts using the XVIVO Heart Preservation System (XHPS) is a safe and effective way to preserve and transport hearts for transplantation.

DETAILED DESCRIPTION:
This is a continuation of the PRESERVE IDE trial to provide additional data evaluating the safety and effectiveness of the XVIVO Heart Assist Transport System. The PRESERVE Continued Access Protocol (CAP) will utilize the XHAT System to preserve donor hearts that may not meet current standard donor heart acceptance criteria with the intention of these hearts being transplanted. The CAP has been implemented to allow patients and physicians access to the XHAT System while a Post-Market Approval (PMA) application is being submitted and reviewed.

ELIGIBILITY:
Inclusion Criteria Recipient:

To be eligible to participate in this study, a recipient must meet all the following criteria:

1. Age ³18 years.
2. Signed informed consent form (ICF).
3. Listed for heart transplantation.

Exclusion Criteria Recipient:

1. Previous solid organ or bone marrow transplantation.
2. Requires a multi-organ transplant.
3. Subject is enrolled and ongoing in another investigational pharmaceutical or medical device clinical trial (Exception: observational studies are permitted).
4. Subject is on mechanical circulatory support pre-transplant other than durable LVAD, Impella or intra-aortic balloon pump (IABP).
5. History of complex congenital heart disease ie: single ventricle physiology (per Investigator's discretion and XVIVO review).
6. Subject on renal replacement therapy/dialysis.
7. Ventilator dependence (subject is intubated at time of transplant/unable to provide consent or re-affirmation of consent).
8. Sensitized participants meeting any of the following:

   * Participant with calculated Panel Reactive Antibody (cPRA) greater than 50%
   * Participant undergoing any desensitization treatment (also with cPRA less than 50%)
   * Participant with a positive prospective crossmatch and/or a positive virtual cross match

Donor Inclusion Criteria:

To be eligible to participate in this study, the donor heart must meet the following criteria:

1. Estimated Cross Clamp Time ≥4 hours OR
2. Estimated Cross Clamp ≥ 2 hours AND

Any one or more of the following:

* Age ≥50 years
* LVEF 40% - 50% at time of provisional acceptance. (Refer to section 6.3.4 for definition of provisional acceptance).
* Down-time ≥20 minutes
* Hypertrophy septal thickness >12 - ≤16mm
* Angiographic luminal irregularities with no significant CAD OR 1) Donation after Circulatory Death (DCD)

Donor Exclusion Criteria:

Donor hearts that meet any of the following criteria will be excluded from transplantation in this study:

1. Unstable hemodynamics requiring high-dose inotropic support.
2. Significantly abnormal coronary angiogram defined as CAD > 50% stenosis of one or more vessels or if the donor heart exhibits any contusions, structural damage, gross abnormalities, or palpable CAD on final examination.
3. Moderate to severe cardiac valve pathology.
4. Investigator's clinical decision to exclude from trial.
5. Previous sternotomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
The percentage of patient treatment success rate | 30 days post transplantation
  The percentage of patient treatment success rate at 30-days post transplantation. The treatment success is defined as freedom from treatment failure.
The percentage of patient survival | Post-operative Day 365.
  The percentage of patient survival at 365 days from the date of transplant. The long-term safety success is defined as survival.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lowe, Study Director — XVIVO Perfusion
Locations (12):
- United States (12):
  - UC San Diego Health, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Washington University - Barnes Jewish Health Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No